CLINICAL TRIAL: NCT00325572
Title: Evaluation and Treatment of Copper/Zinc Imbalance in Children With Autism
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy to proceed to Phase 2
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Jeanette C. Ramer, Professor of Pediatrics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23275
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-05

CONDITIONS: Autism; Pervasive Developmental Disorder
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral zinc and vitamin C supplementation (Active Comparator): Participant will receive oral zinc and vitamin C supplementation based on the child's weight. Blood levels of zinc, copper, liver and renal function as well as blood counts will be measured. Copper to zinc ratio will be calculated at 6 and 16 weeks
  Interventions: Drug: oral zinc and vitamin C supplements
- Oral Placebo (Placebo Comparator): Participant will receive placebo liquid with volume based on child's weight to match the amount given to participants in the experimental group.
  Interventions: Other: oral Placebo

INTERVENTIONS:
Drug: oral zinc and vitamin C supplements — Each child will be provided separate suspensions containing zinc and vitamin C to be taken twice per day. The dose will be based on the child's weight and be titrated by checking copper/zinc ratio at 6 weeks of treatment. Monitoring of liver, renal functions and CBC will occur at the end of supplementation
  Arms: Oral zinc and vitamin C supplementation
Other: oral Placebo — Each child will be provided separate Placebo suspensions C to be taken twice per day. The dose will be based on the child's weight and be titrated by checking copper/zinc ratio at 6 weeks of treatment. Monitoring of liver, renal functions and CBC will occur at the end of supplementation
  Arms: Oral Placebo

SUMMARY:
There are two phases to the study. The first will examine serum copper and zinc levels and copper/zinc ratio in children (ages 3-8) who have autism and compare them to levels from same sex and age children who are developing typically. The hypothesis is that there is a significant difference in the copper/zinc ratio between young children who have autism and their typically developing peers.

The second phase of the study will evaluate the effect of dietary supplementation using zinc and vitamin C for 16 weeks on selected symptoms of autism. Children with autism will be enrolled on the basis of copper/zinc ratios greater than 2.0, and as determined to be statistically higher than typically developing children. Measurements of serum copper, zinc and unbound copper will be obtained prior to, at the mid-point and end of the trial. Those children whose ratios have not fallen below 1.25, the top of the currently recognized range will have the zinc and vitamin C doses adjusted for the duration of the trial. Detailed evaluation of language skills, and a variety of behaviors will be evaluated prior to and after supplementation. The study will be placebo-controlled and double blind. Those children enrolled in the placebo arm will be offered a full trial of supplements at the end of the their participation in the study.

The hypothesis to be tested is whether correction of elevated copper to zinc ratios in children with autism can be accomplished by oral supplementation with zinc and vitamin C and if these children show measurable and significant changes in receptive or expressive language or behavioral parameters associated with autism.

ELIGIBILITY:
Inclusion Criteria:

* Ages 3-8 years
* Diagnosis of autism spectrum disorder
* Serum copper/zinc ratio greater than 2.0 or as determined in phase 1 of the study

Exclusion Criteria:

* Known chromosomal disorder or neurological disorders other than autism

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2006-11; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette C Ramer, MD, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Penn State Children's Hospital, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was begun in January, 2006. The participants were recruited from a developmental pediatrics outpatient clinic and comparison patients were recruited from a general pediatrics clinic and an allergy clinic.
Pre-assignment Details: The Modified Checklist for Autism in Toddlers and the Social Responsiveness Scale were used as screens. 3 children were excluded from the comparison group because of scores outside the typical range. 4 children were excluded from the autism study group because they failed to meet criteria for autism using the Autism Diagnostic Interview-Revised.
Groups:
- Zinc and Vitamin C Supplementation: Participant will receive oral zinc and vitamin C supplementation based on the child's weight. Blood levels of zinc, copper, liver and renal function as well as blood counts will be measured. Copper to zinc ratio will be calculated at 6 and 16 weeks
- Placebo Group: Participant will receive placebo liquid with volume based on child's weight to match the amount given to participants in the experimental group.
Period: PHASE I
Arm/Group | Zinc and Vitamin C Supplementation | Placebo Group
Started | 45 | 44
Completed | 45 | 44
Not Completed | 0 | 0
Period: PHASE ii
Arm/Group | Zinc and Vitamin C Supplementation | Placebo Group
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zinc and Vitamin C Supplementation | Placebo Group | Total
Number analyzed (Participants) | 45 | 44 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 45 | 44 | 89
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.5 (1.2) | 5.9 (1.9) | 5.12 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 21 | 25
  Male | 41 | 23 | 64
Region of Enrollment [Number; unit: participants]
  United States | 45 | 44 | 89

OUTCOME MEASURES:

1. Primary Outcome: Copper/Zinc Ratio of Children With Autism Compared to Typically Developing Children Phase 2: Change in Copper/Zinc Ratio With Supplementation of Zinc and Vitamin C
Description: Phase 2 was not initiated; no data was collected.
Time Frame: 16 weeks
Population: Phase 2 was not initiated; no data was collected.
Arm/Group | Zinc and Vitamin C Supplementation | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were monitored / assessed for Phase 1 of the study.
Arm/Group | Zinc and Vitamin C Supplementation | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 0/45 | 0/44

LIMITATIONS AND CAVEATS:
Trial was not completed and did not progress past Phase 1 of the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes